CLINICAL TRIAL: NCT05310838
Title: Optimizing Engagement in Services for First-Episode Psychosis (FEP) in the Community Mental Health Setting
Brief Title: Optimizing Engagement in Services for First-Episode Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, San Bernardino (Other)
Collaborators: University of Southern California (Other); Olive View-UCLA Education & Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Maria Santos, Assistant Professor, California State University, San Bernardino
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY2020-167; K23MH119313 (NIH)
Record Dates: First submitted 2022-02-10; First posted 2022-04-05 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Engagement, Patient; First Episode Psychosis
Keywords: First Episode Psychosis; Behavioral Activation; Engagement; Latinx
MeSH Terms: conditions — Patient Participation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation for First Episode Psychosis (Experimental): Patients will receive BA for FEP in individual session format provided by the PI based on a manual adapted for this study.
  Interventions: Behavioral: Behavioral Activation for First Episode Psychosis
- Treatment at Usual (Active Comparator): Patients randomized to TAU will receive typical clinic care offered beyond psychiatric services.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Behavioral Activation for First Episode Psychosis — Sessions will be offered weekly and dyads can complete the intervention during a 6-month period to accommodate competing demands encountered by the population.
  Arms: Behavioral Activation for First Episode Psychosis
Behavioral: Treatment As Usual — Given this condition, patients may also receive individual rehabilitation and/or group psychosocial interventions as part of typical clinic care.
  Arms: Treatment at Usual

SUMMARY:
This study will compare a 12-session behavioral activation (BA) intervention modified for first-episode psychosis (FEP) to usual community mental health care (i.e., treatment-as-usual; TAU) delivered over 6 months with a sample of Latinos with FEP and their families. Comparable family group sessions will also be delivered to participants in both conditions. It is expected that BA participants will show better engagement than TAU participants.

DETAILED DESCRIPTION:
After an initial pre-screen, screening, and pre-intervention assessment, enrolled participants will be randomized to either BA or TAU. The study intervention phase will last up to 6 months, during which time BA participants will receive up to 12 one-on-one BA sessions and TAU participants will receive the usual care (e.g., medication management and any other service [e.g., group counseling]). Participants will be assessed at post-intervention, 1-month-post-intervention, and 6-month-post-intervention. The primary objective of aim 1 is to examine whether BA for FEP improves engagement in services better than TAU among Latinos with FEP and their families. Secondary objectives of aim 1 are to examine whether BA participants show greater improvements in quality of life, symptoms (e.g., psychosis, depression), functioning, and recovery compared to TAU participants, and whether BA participants have greater remission rates than the TAU group at 1- and 6-month post-intervention. Additionally, the association between potential BA mediators and engagement will be examined to identify mechanisms of engagement. Potential predictors of engagement will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as Latino
* Age 15 to 35
* Diagnostic & Statistical Manual of Mental Disorders-5 diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, brief psychotic disorder, other specified schizophrenia spectrum, affective psychosis, and other psychotic disorder criteria
* Ability to speak English or Spanish
* Caregiver willing to consent to participate in the study and care
* Ability to provide fully informed consent

Exclusion Criteria:

* Diagnosis of psychotic disorder due to another medical condition or substance/medication-induced psychotic disorder
* Presence of a serious medical condition
* 3≤ years after the onset

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Engagement on the Patient Activation Measure (PAM13) at Post-Intervention | Change from Pre-intervention PAM13 at Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  PAM13 is a 13-item self-report short form of a patient's engagement in the care process at four stages. PAM13 shows high reliability that is stable across chronic illnesses and high construct validity, and measures change over time. Items are rated on a 4-point Likert scale (totally disagree to totally agree) with higher scores reflecting higher activation; respondent may select 'not applicable.'
Change in Engagement on the Patient Activation Measure (PAM13) at 1-Month Post-Intervention | Change from Pre-intervention PAM13 at 1-month-post-intervention
  PAM13 is a 13-item self-report short form of a patient's engagement in the care process at four stages. PAM13 shows high reliability that is stable across chronic illnesses and high construct validity, and measures change over time. Items are rated on a 4-point Likert scale (totally disagree to totally agree) with higher scores reflecting higher activation; respondent may select 'not applicable.'
Change in Engagement on the Patient Activation Measure (PAM13) at 6-Months Post-Intervention | Change from Pre-intervention PAM13 at 6-months-post-intervention
  PAM13 is a 13-item self-report short form of a patient's engagement in the care process at four stages. PAM13 shows high reliability that is stable across chronic illnesses and high construct validity, and measures change over time. Items are rated on a 4-point Likert scale (totally disagree to totally agree) with higher scores reflecting higher activation; respondent may select 'not applicable.'
Engagement as measured by the Service Engagement Scale (SES) | Weekly per session up to 12 sessions, up to 6 months
  The 14-item provider rated SES has demonstrated good reliability and validity and reflects client availability, collaboration, help-seeking, and adherence. Items are rated on a 4-point Likert scale with higher scores reflecting clients' greater levels of difficulty engaging with services. The SES is a secondary measure of service engagement.

SECONDARY OUTCOMES:
Change in Quality of Life on the Heinrichs-Carpenter Quality of Life Scale (QLS) at Post-Intervention | Change from Pre-intervention QLS at Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  The QLS is a 21-item, clinician-administered, semi-structured interview on a 7-point scale with higher scores reflecting normal or unimpaired functioning. It has shown high sensitivity to change and treatment effect. The total score is the main secondary outcome of interest.
Change in Quality of Life on the Heinrichs-Carpenter Quality of Life Scale (QLS) at 1-Month Post-Intervention | Change from Pre-intervention QLS at 1-month-post-intervention
  The QLS is a 21-item, clinician-administered, semi-structured interview on a 7-point scale with higher scores reflecting normal or unimpaired functioning. It has shown high sensitivity to change and treatment effect. The total score is the main secondary outcome of interest.
Change in Quality of Life on the Heinrichs-Carpenter Quality of Life Scale (QLS) at 6-Months Post-Intervention | Change from Pre-intervention QLS at 6-months-post-intervention
  The QLS is a 21-item, clinician-administered, semi-structured interview on a 7-point scale with higher scores reflecting normal or unimpaired functioning. It has shown high sensitivity to change and treatment effect. The total score is the main secondary outcome of interest.
Change in Quality of Life on the Modified Lehman Quality of Life Inventory (QOLI-M) at Post-Intervention | Change from Pre-intervention QOLI-M at Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  The QOLI-M has well established psychometric properties with individuals with serious mental illness (SMI) and will be used to derive overall subjective quality of life and objective and subjective quality of social and family interaction ratings. The QOLI-M, not the QLS, assesses general quality of life which focuses on areas beyond those affected by psychotic illness.
Change in Quality of Life on the Modified Lehman Quality of Life Inventory (QOLI-M) at 1-Month Post-Intervention | Change from Pre-intervention QOLI-M at 1-month-post-intervention
  The QOLI-M has well established psychometric properties with individuals with serious mental illness (SMI) and will be used to derive overall subjective quality of life and objective and subjective quality of social and family interaction ratings. The QOLI-M, not the QLS, assesses general quality of life which focuses on areas beyond those affected by psychotic illness.
Change in Quality of Life on the Modified Lehman Quality of Life Inventory (QOLI-M) at 6-Months Post-Intervention | Change from Pre-intervention QOLI-M at at 6-months-post-intervention
  The QOLI-M has well established psychometric properties with individuals with serious mental illness (SMI) and will be used to derive overall subjective quality of life and objective and subjective quality of social and family interaction ratings. The QOLI-M, not the QLS, assesses general quality of life which focuses on areas beyond those affected by psychotic illness.
Change in Symptoms on the Positive And Negative Syndrome Scale (PANSS) at Post-Intervention | Change from Pre-intervention PANSS at Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  This 30-item widely-used clinician-administered instrument measures psychosis symptom severity and remission. Scores 4 ≤ on delusions, conceptual disorganization, hallucinatory behavior, mannerisms & posturing, and unusual thought content will be considered in remission.
Change in Symptoms on the Positive And Negative Syndrome Scale (PANSS) at 1-Month Post-Intervention | Change from Pre-intervention PANSS at 1-month-post-intervention
  This 30-item widely-used clinician-administered instrument measures psychosis symptom severity and remission. Scores 4 ≤ on delusions, conceptual disorganization, hallucinatory behavior, mannerisms & posturing, and unusual thought content will be considered in remission.
Change in Symptoms on the Positive And Negative Syndrome Scale (PANSS) at 6-Months Post-Intervention | Change from Pre-intervention PANSS at 6-months-post-intervention
  This 30-item widely-used clinician-administered instrument measures psychosis symptom severity and remission. Scores 4 ≤ on delusions, conceptual disorganization, hallucinatory behavior, mannerisms & posturing, and unusual thought content will be considered in remission.
Change in Functioning on the Strauss-Carpenter level of Function Scale (Strauss-Carpenter) at Post-Intervention | Change from Pre-intervention Strauss-Carpenter at Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  The Strauss-Carpenter is a semi-structured interviewer-administered scale that assesses functioning in social contacts, work, symptomatology, and function. Items are rated on a five-point scale (0-4) with higher scores reflecting better functioning.
Change in Functioning on the Strauss-Carpenter level of Function Scale (Strauss-Carpenter) at 1-Month Post-Intervention | Change from Pre-intervention Strauss-Carpenter at 1-month-post-intervention
  The Strauss-Carpenter is a semi-structured interviewer-administered scale that assesses functioning in social contacts, work, symptomatology, and function. Items are rated on a five-point scale (0-4) with higher scores reflecting better functioning.
Change in Functioning on the Strauss-Carpenter level of Function Scale (Strauss-Carpenter) at 6-Months Post-Intervention | Change from Pre-intervention Strauss-Carpenter at 6-months-post-intervention
  The Strauss-Carpenter is a semi-structured interviewer-administered scale that assesses functioning in social contacts, work, symptomatology, and function. Items are rated on a five-point scale (0-4) with higher scores reflecting better functioning.
Change in Depression on the Calgary Depression Scale (CDS) at Post-Intervention | Change from Pre-intervention CDS at Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  The CDS is an interview-based 9-item scale that measures depression severity in people with schizophrenia and is valid and reliable. Items are rated on a four-point scale with higher scores reflecting greater severity of symptoms.
Change in Depression on the Calgary Depression Scale (CDS) at 1-Month Post-Intervention | Change from Pre-intervention CDS at 1-month-post-intervention
  The CDS is an interview-based 9-item scale that measures depression severity in people with schizophrenia and is valid and reliable. Items are rated on a four-point scale with higher scores reflecting greater severity of symptoms.
Change in Depression on the Calgary Depression Scale (CDS) at 6-Months Post-Intervention | Change from Pre-intervention CDS at 6-months-post-intervention
  The CDS is an interview-based 9-item scale that measures depression severity in people with schizophrenia and is valid and reliable. Items are rated on a four-point scale with higher scores reflecting greater severity of symptoms.
Change in Recovery as measured by the Maryland Assessment of Recovery in People with SMI (MARS) at Post-Intervention | Change from Pre-intervention MARS at Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  The 25-item patient-report MARS measures recovery and has excellent internal consistency and test-retest reliability and good face and content validity. Items are rated on a five-point scale with higher scores reflecting greater self-reported recovery.
Change in Recovery as measured by the Maryland Assessment of Recovery in People with SMI (MARS) at 1-Month Post-Intervention | Change from Pre-intervention MARS at 1-month-post-intervention
  The 25-item patient-report MARS measures recovery and has excellent internal consistency and test-retest reliability and good face and content validity. Items are rated on a five-point scale with higher scores reflecting greater self-reported recovery.
Change in Recovery as measured by the Maryland Assessment of Recovery in People with SMI (MARS) at 6-Months Post-Intervention | Change from Pre-intervention MARS at 6-months-post-intervention
  The 25-item patient-report MARS measures recovery and has excellent internal consistency and test-retest reliability and good face and content validity. Items are rated on a five-point scale with higher scores reflecting greater self-reported recovery.
PANSS-based Remission Rates at Post-Intervention | Remission at Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  Scores 4 ≤ on delusions, conceptual disorganization, hallucinatory behavior, mannerisms & posturing, and unusual thought content will be considered in remission.
PANSS-based Remission Rates at 1-Month Post-Intervention | Remission at 1-month-post-intervention
  Scores 4 ≤ on delusions, conceptual disorganization, hallucinatory behavior, mannerisms & posturing, and unusual thought content will be considered in remission.
PANSS-based Remission Rates at 6-Months Post-Intervention | Remission at 6-months-post-intervention
  Scores 4 ≤ on delusions, conceptual disorganization, hallucinatory behavior, mannerisms & posturing, and unusual thought content will be considered in remission.

OTHER OUTCOMES:
Change in Activation as measured by the Behavioral Activation for Depression Scale-Short Form (BADS-SF) at Post-Intervention | Change from Pre-intervention BADS-SF at Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  The 9-item self-report BADS-SF tracks when and how changes in activation occur (7-point scale; not at all to completely). It has shown good internal consistency reliability, construct validity, and predictive validity. BADS-SF is the primary measure of activation.
Change in Activation as measured by the Behavioral Activation for Depression Scale-Short Form (BADS-SF) at 1-Month Post-Intervention | Change from Pre-intervention BADS-SF at 1-month-post-intervention
  The 9-item self-report BADS-SF tracks when and how changes in activation occur (7-point scale; not at all to completely). It has shown good internal consistency reliability, construct validity, and predictive validity. BADS-SF is the primary measure of activation.
Change in Activation as measured by the Behavioral Activation for Depression Scale-Short Form (BADS-SF) at 6-Months Post-Intervention | Change from Pre-intervention BADS-SF at 6-months-post-intervention
  The 9-item self-report BADS-SF tracks when and how changes in activation occur (7-point scale; not at all to completely). It has shown good internal consistency reliability, construct validity, and predictive validity. BADS-SF is the primary measure of activation.
Activation as measured by the Behavioral Activation Homework Completion Observer-Based Coding System (BA HC) | Weekly per session up to 12 sessions, up to 6 months
  BA HC permits reliable coding of the characterization and completion of BA homework, including type of assignment, realm of functioning it targets, and the extent of homework completion. It will be used as a secondary measure of activation for BA.
Change in Environmental Reward as measured by the Reward Probability Index (RPI) at Post-Intervention | Change from Pre-intervention RPI at Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  RPI is a 20-item self-report measure of contact with environmental reward, which is theorized to maintain healthy behavior per behavioral models of psychopathology, with good internal consistency, test-retest reliability, and discriminant, predictive, and convergent validity. Items are rated on a 4-point Likert scale with higher scores indicating higher levels of reinforcement.
Change in Environmental Reward as measured by the Reward Probability Index (RPI) at 1-Month Post-Intervention | Change from Pre-intervention RPI at 1-month-post-intervention
  RPI is a 20-item self-report measure of contact with environmental reward, which is theorized to maintain healthy behavior per behavioral models of psychopathology, with good internal consistency, test-retest reliability, and discriminant, predictive, and convergent validity. Items are rated on a 4-point Likert scale with higher scores indicating higher levels of reinforcement.
Change in Environmental Reward as measured by the Reward Probability Index (RPI) at 6-Months Post-Intervention | Change from Pre-intervention RPI at 6-months-post-intervention
  RPI is a 20-item self-report measure of contact with environmental reward, which is theorized to maintain healthy behavior per behavioral models of psychopathology, with good internal consistency, test-retest reliability, and discriminant, predictive, and convergent validity. Items are rated on a 4-point Likert scale with higher scores indicating higher levels of reinforcement.
Change in medication adherence as measured by the Brief Adherence Rating Scale (BARS) at Post-Intervention | Change from Pre-intervention BARS at Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  The 4-item BARS is a brief, clinician-administered instrument to assess oral antipsychotic medication adherence and has good sensitivity (73%) and specificity (74%) in identifying non-adherent outpatients (defined as <70% mean electronic monitoring adherence).
Change in medication adherence as measured by the Brief Adherence Rating Scale (BARS) at 1-Month Post-Intervention | Change from Pre-intervention BARS at 1-month-post-intervention
  The 4-item BARS is a brief, clinician-administered instrument to assess oral antipsychotic medication adherence and has good sensitivity (73%) and specificity (74%) in identifying non-adherent outpatients (defined as <70% mean electronic monitoring adherence).
Change in medication adherence as measured by the Brief Adherence Rating Scale (BARS) at 6-Months Post-Intervention | Change from Pre-intervention BARS at 6-months-post-intervention
  The 4-item BARS is a brief, clinician-administered instrument to assess oral antipsychotic medication adherence and has good sensitivity (73%) and specificity (74%) in identifying non-adherent outpatients (defined as <70% mean electronic monitoring adherence).
Alliance as measured by the Working Alliance Inventory - Short Form (WAI-SF) | Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  The 12-item WAI-SF measures agreement on goals and tasks of therapy and the bond between the therapist and the client and has demonstrated good reliability and convergent validity. Items are rated on a 5-point Likert scale with higher scores indicating a better therapeutic alliance. The WAI-SF will be used to assess the patient-provider alliance.
Person-centered care as measured by the Combined Assessment of Psychiatric Environments (CAPE) | Post-intervention (after 12th session or 6-months after start of intervention, whichever comes first)
  CAPE assesses patient perspective patient-centered care and shows internal consistency reliability, test-retest reliability, and construct and criterion validity.
Family involvement | Weekly per session up to 12 sessions, up to 6 months
  Family involvement, or whether a family member was present at a service encounter, will be assessed by an independent observer based on review of service. This method has been used in prior early intervention studies.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Santos, PhD, Principal Investigator — California State University, San Bernardino
Locations (2):
- United States (2):
  - San Fernando Mental Health Center, Granada Hills, California
  - Olive View - UCLA Medical Center, Sylmar, California

IPD SHARING:
Plan to Share IPD: No